CLINICAL TRIAL: NCT03641820
Title: Correlative Factors of Cognitive Dysfunction in Patients With Cancer Pain: a Cross-sectional Study From China
Brief Title: Cognitive Dysfunction in Patients With Cancer Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FJZL20180407
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the occurrence of cognitive dysfunction in cancer patients with pain in China.Analysis of patients with different cancer pain, different analgesic drugs and different treatments are associated with the severity of cognitive dysfunction, to provide relevant evidence for the next screening, prediction, prevention and treatment. In order to achieve the purpose of improving the quality of life of cancer patients.

DETAILED DESCRIPTION:
Cross-sectional survey in patients with cancer pain is used in the outpatient clinics and wards of five cancer hospitals in China.

This study is to survey the incidence of cognitive dysfunction in Chinese cancer patients, and the related factors of cognitive dysfunction, demographic characteristics (economic situation, education, gender, age), disease status (tumor type, staging) ), analgesic treatment (NRS score, with or without analgesic drugs, analgesic drug name, dose), anti-tumor treatment (with or without anti-tumor treatment, surgery, radiotherapy, chemotherapy, time interval from last treatment, chemotherapy drugs) and so on.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor patient with pain are confirmed by histopathology or cytology (NRS score ≥ 1);
* Understand Chinese through verbal and written communication, read and write Chinese, numbers, and complete questionnaire surveys;
* Male or female, age 18-75 years old;
* ECOG 0-2, expected to survive for more than 3 months;
* no obvious dysfunction of heart, lung, liver, kidney, blood system (≤I degree);
* patients voluntarily sign informed consent

Exclusion Criteria:

* Pregnant women and lactating women.
* Also participate in clinical trials of drugs that have not been approved for marketing.
* Patients with depression (evaluated by the Hamilton Depression Scale).
* Active bleeding or bleeding tendency.
* Serious or uncontrolled medical conditions and infected people.
* Patients with structural heart disease, such as coronary heart disease, unstable angina, especially patients with congestive heart failure and atrial fibrillation, atrial flutter history, and patients with hypertension, hypercoagulable state and severe cerebrovascular disease.
* History of thromboembolic disease; long-term oral administration of aspirin and other anticoagulants.
* Preventive Whole Brain Irradiation (PCI).
* Bone marrow invasion or bone marrow metastasis.
* Patients with severe or uncontrollable mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant tumor patient with pain
Sampling Method: Probability Sample
Enrollment: 928 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Cancer-related cognitive dysfunction patient with pain | 6 months
  Statistical analysis was performed SPSS 21.0. The t test was used for comparison between groups, and the X2 test was used for the count data. The logistic regression model was used for multivariate analysis. The regression coefficient, P value and OR value were calculated by age, ethnicity, education level, treatment plan and income as covariates.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nursing, Fujian Provincial Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided